CLINICAL TRIAL: NCT03452306
Title: Four-way Crossover, Open-label, Single-dose, Bioequivalence Study of Metformin (LLC "GEROPHARM", Russia) 750 mg Tablets Extended Release Versus Glucophage® Long (Merck Santé S.A.S, France) 750 mg Tablets Extended Release in Normal Healthy Subjects Under Fasting and Fed Conditions
Brief Title: Bioequivalence Study of Metformin 750 mg Tablets XR Versus Glucophage® Long 750 mg Tablets XR In Normal Healthy Subjects Under Fasting and Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Geropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BIOMET-LONG
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Bioequivalence
Keywords: AUC; Cmax; Pharmacokinetics; metformin; fed; fasting
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency; Fasting | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: four-way crossover
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): First aIntervention Period:
  Single administered dose of Metformin (750 mg tablet extended-release in a fasting condition
  Third Intervention Period:
  Single administered dose of Metformin (750 mg tablet extended-release) in a fed condition
  Interventions: Drug: Metformine; Drug: Metformin
- Glucophage® Long (Active Comparator): Second Intervention Period:
  Single administered dose of Glucophage® ( 750 mg tablet extended-release) in a fasting condition
  Fourth Intervention Period:
  Single administered dose of Glucophage® ( 750 mg tablet extended-release) in a fed condition
  Interventions: Drug: Glucophage® Long

INTERVENTIONS:
Drug: Metformine — First aIntervention Period:
  Single administered dose of Metformin (750 mg tablet extended-release) in a fasting condition
  Other Names: fasting condition
  Arms: Metformin
Drug: Glucophage® Long — Second Intervention Period:
  Single administered dose of Glucophage® (750 mg tablet extended-release) in a fasting condition
  Other Names: fasting condition
  Arms: Glucophage® Long
Drug: Metformin — Third Intervention Period:
  Single administered dose of Metformin (750 mg tablet extended-release) in a fed condition
  Other Names: fed condition
  Arms: Metformin
Drug: Glucophage® Long — Fourth Intervention Period:
  Single administered dose of Metformin (750 mg tablet extended-release) in a fed condition
  Other Names: fed condition
  Arms: Glucophage® Long

SUMMARY:
Bioequivalence Study of 2 formulation of metformin (Metformin GEROPHARM vers. Glucophage® Long Merck )

DETAILED DESCRIPTION:
Study to evaluate the bioequivalence of orally administered metformin preparations, Extended release tablets, 750 mg in normal healthy subjects under fasting and fed conditions

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Healthy male and female subjects aged 18 to 45 years.
* Verified diagnosis is "healthy" according to data Standard clinical, laboratory and Instrumental methods of examination.
* Have a body mass index between 18,5 and 27 kg/m2.
* Females must have a negative pregnancy test.
* Subjects must use, with their partner, methods of highly effective contraception throughout the study and 30 days after the end of study.

Exclusion Criteria:

* History of serious allergic problems/events
* Medicinal intolerance.
* History of allergic reactions to memantine or investigator's product components
* Any acute and chronic diseases of the cardiovascular system, cardiovascular, bronchopulmonary, neuroendocrine systems, as well as diseases of the gastrointestinal tract, liver, kidneys, blood.
* Acute infectious diseases in less than 4 weeks before the start of the study.
* Subjects who have taken medication 4 weeks preceding before the study.
* Subjects who have taken any drugs known effects on hemodynamics or to induce or inhibit hepatic drug metabolism within 30 days prior to administration of the study medication (examples of inducers: barbiturates, omeprazole, etc.).
* Donation of plasma (450 mL or more) within 2 month prior to administration of the study medication.
* History of significant alcohol or drugs abuse or any indication of the regular use of more than 10 units of alcohol per week (1 Unit = 200 mL of wine or 500 mL of beer or 50 mL of alcohol 40%).
* Smokers.
* Participation in other clinical training is less than than for 3 months before the study.
* Lack of signed informed consent form.
* ECG or vital signs abnormalities (clinically significant).
* Positive testing for alcohol, drugs, pregnancy.
* Dehydration due to diarrhea, vomiting, or other causes within the last 24 hours before the start of the study.
* Any diet, for example, vegetarian, for 2 weeks before taking the study medications.
* Women with preserved reproductive potential who have unprotected sexual intercourse with an unsterilized male partner within 30 days prior to taking the study medication.
* Heart rate below 60 or above 80 beats per minute.
* Systolic blood pressure less than 110 mm Hg or more than 139 mm Hg.
* Diastolic blood pressure less than 70 mm Hg or more than 89 mm Hg.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-07-22 (Actual); Study Completion 2017-07-22 (Actual)

PRIMARY OUTCOMES:
Cmax | 0 hours (pre-dose), as well as at 0.5, 1.0, 2.0, 3.0, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 8.0, 9.0, 10.0, 12.0, 16.0, 20.0, 24.0, 30.0 and 36 hours post-dose
  Pharmacokinetics of metformin by Assessment of Observed Maximum Plasma Concentration (Cmax)
AUC(0-t) | 0 hours (pre-dose), as well as at 0.5, 1.0, 2.0, 3.0, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 8.0, 9.0, 10.0, 12.0, 16.0, 20.0, 24.0, 30.0 and 36 hours post-dose
  Pharmacokinetics of metformin by Assessment of Area Under the Curve From Time Zero Extrapolated to "t" (AUC(0-t))

CONTACTS AND LOCATIONS:
Locations (1):
- Yarosslavl Clinical Hospital #3, Yaroslavl, Russia

IPD SHARING:
Plan to Share IPD: No